CLINICAL TRIAL: NCT06597227
Title: Comparison of Clinical Efficacy of Proximal Gastrectomy Vs Total Gastrectomy in Locally Advanced Upper Gastric Cancer After SOX Combined with Anti-PD-1 Neoadjuvant Therapy：a Prospective, Multi-center, Randomised，controlled Trial
Brief Title: Proximal Gastrectomy Vs Total Gastrectomy in Locally Advanced Upper Gastric Cancer After Neoadjuvant Therapy
Acronym: TJHGC01
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Guihua Wang (Other)
Collaborators: Fudan University (Other); Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); The First Affiliated Hospital of Air Force Medicial University (Other); Xiangya Hospital of Central South University (Other); Shandong First Medical University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); The First Medical Center of Chinese PLA General Hospital (Other); Affiliated Hospital of Qinghai University (Other); Qilu Hospital of Shandong University (Other); Ruijin Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Southern Medical University, China (Other); Zhongnan Hospital (Other); Shanxi Bethune Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Fujian Medical University Union Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Jingzhou Central Hospital (Other); Xiangyang Central Hospital (Other); Yichang Central People's Hospital (Other); People's Hospital of Macheng City (Unknown); The First Affiliated Hospital of University of South China (Other)
Responsible Party: Sponsor-Investigator, Guihua Wang, Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-S029
Record Dates: First submitted 2024-09-05; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Locally Advanced Gastric Cancer
Keywords: Locally advanced gastric cancer; neoadjuvant chemotherapy; immunotherapy; Proximal radical gastrectomy; total radical gastrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Proximal radical gastrectomy group (Experimental): Patients with locally advanced upper gastric cancer were enrolled for 4 cycles of SOX combined with anti-PD-1 neoadjuvant therapy. After the completion of neoadjuvant therapy, the efficacy was evaluated, and the patients were divided into two groups according to the remission of lesions: (1) PD (Progressive disease) and SD (Stable disease) patients were replaced with conservative treatment or surgical treatment after MDT (Multi-disciplinary Treatment) discussion; (2) For PR (Partial response) and CCR (Clinical complete response) patients, if the patients met the criteria for proximal gastric radical surgery, the enrolled patients were randomly divided into 2 cohorts, which were divided into experimental group : the group of proximal gastric radical surgery; Four cycles of SOX combined with anti-PD-1 adjuvant therapy continued after surgery, and anti-PD-1 adjuvant therapy lasted for 1 year.
  Interventions: Procedure: Proximal radical gastrectomy
- Total radical gastrectomy group (Active Comparator): Patients with untreated, operable locally advanced upper gastric cancer who signed informed consent and met the screening criteria were enrolled for 4 cycles of SOX combined with anti-PD-1 neoadjuvant therapy. After the completion of neoadjuvant therapy, the efficacy was evaluated, and the patients were divided into two groups according to the remission of lesions: (1) PD and SD patients were replaced with conservative treatment or surgical treatment after MDT discussion; (2) For PR and CCR patients, if the patients met the criteria for proximal gastric radical surgery, the enrolled patients were randomly divided into 2 cohorts, Cohort 2 (control group) : total radical gastrectomy group. Four cycles of SOX combined with anti-PD-1 adjuvant therapy continued after surgery, and anti-PD-1 adjuvant therapy lasted for 1 year.
  Interventions: Procedure: Total radical gastrectomy

INTERVENTIONS:
Procedure: Proximal radical gastrectomy — Proximal radical gastrectomy : Dissection of lymph nodes No.1,2,3a,4sa,4sb,7,8a, 9, 11p, 11dare recommended. The tumor involved more than 3cm of esophagus and additional dissection No.19, 20, 110. Gastrointestinal reconstruction method: double channel anastomosis is recommended, and other anastomosis methods can be carried out according to the surgeon's habit.
  Arms: Proximal radical gastrectomy group
Procedure: Total radical gastrectomy — total radical gastrectomy : Dissection of lymph nodes No.1-7, 8a, 9, 11p, 11d, 12a are recommended. The tumor involved more than 3cm of esophagus and additional dissection No.19, 20, 110. Gastrointestinal reconstruction method: Roux⁃en⁃Y anastomosis is recommended
  Arms: Total radical gastrectomy group

SUMMARY:
We plan to evaluate the efficacy and safety of proximal gastric vs. total gastric radical resection after SOX combined with anti-PD-1 neoadjuvant therapy in locally advanced upper gastric cancer

DETAILED DESCRIPTION:
Gastric cancer is one of the most common malignant tumors in China, and its morbidity and mortality rank among the top three for a long time.How to improve the survival rate of patients with advanced gastric cancer is the key to improve the prognosis.At present, neoadjuvant chemotherapy combined with immunosuppressants has a higher pathologic complete response (pCR) rate, reduce the clinical stage of tumors and improve the resection rate of radical surgery.Some studies have suggested that preserving partial gastric lymph nodes may enhance immunotherapy efficacy.Proximal radical gastrectomy versus total radical gastrectomy can reduce the scope of surgical resection and preserve some lymph nodes, which may contribute to long-term survival and improve postoperative quality of life of patients. It is expected to translate the short-term benefit of neoadjuvant immunotherapy into the benefit of patient overall survival (OS) rate.At the same time, our previous studies have shown that the methylation level of PD-L1 K162 can be used as a new indicator to predict the sensitivity of anti-PD -(L)1 immunotherapy, which is expected to be further confirmed in this clinical trial.Therefore, we plan to conduct a comparative study on the effectiveness and safety of proximal gastric vs. total gastric radical resection after SOX combined with anti-PD-1 neoadjuvant therapy for locally advanced upper gastric cancer, which is expected to propose new changes in surgical methods for gastric cancer and a new indicator for screening the advantages of gastric cancer immunotherapy in the era of immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible to participate in this study, all patients must meet all the following criteria:

  1. The subjects voluntarily joined the study and were able to sign the informed consent with good compliance;
  2. Age 18-75 years old (at the time of signing the informed consent), both male and female;
  3. Histologically and/or cytologically confirmed upper gastric carcinoma (adenocarcinoma), locally advanced according to AJCC Edition 8 criteria, cT3-4 or N+M0 according to endoscopic ultrasound or enhanced CT/MRI scanning (combined with diagnostic laparoscopic exploration if necessary) , and consent to neoadjuvant therapy. Investigators assessed the lesion as resectable or potentially resectable;
  4. Have not received systematic treatment for the current disease, including anti-tumor chemoradiotherapy/immunotherapy;
  5. ECOG score 0-1;
  6. Expected survival ≥6 months;
  7. Preoperative chest, abdominal, pelvic CT or PET-CT to exclude distant metastasis;
  8. The major organs function well and meet the following criteria:

  <!-- -->

  1. Blood routine examination (no blood transfusion within 14 days, no hematopoietic stimulating drugs to correct the state) : hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet (PLT) ≥80×109/L;
  2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Serum total bilirubin (TBIL) ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥60mL/min;
  3. Coagulation function: activated partial thromboplastin time (APTT), International standardized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
  4. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥50%;
  5. Assessed with adequate organ function by doctors. 9. Fertile subjects must use appropriate methods of contraception during the study period and within 120 days after the end of the study, have a negative serological pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects.

Exclusion Criteria:

* To be eligible to participate in this study, all patients must meet all the following criteria:

  1. The subjects voluntarily joined the study and were able to sign the informed consent with good compliance;
  2. Age 18-75 years old (at the time of signing the informed consent), both male and female;
  3. Histologically and/or cytologically confirmed upper gastric carcinoma (adenocarcinoma), locally advanced according to AJCC Edition 8 criteria, cT3-4 or N+M0 according to endoscopic ultrasound or enhanced CT/MRI scanning (combined with diagnostic laparoscopic exploration if necessary) , and consent to neoadjuvant therapy. Investigators assessed the lesion as resectable or potentially resectable;
  4. Have not received systematic treatment for the current disease, including anti-tumor chemoradiotherapy/immunotherapy;
  5. ECOG score 0-1;
  6. Expected survival ≥6 months;
  7. Preoperative chest, abdominal, pelvic CT or PET-CT to exclude distant metastasis;
  8. The major organs function well and meet the following criteria:

  <!-- -->

  1. Blood routine examination (no blood transfusion within 14 days, no hematopoietic stimulating drugs to correct the state) : hemoglobin (Hb) ≥90g/L; Absolute neutrophil count (ANC) ≥1.5×109/L; Platelet (PLT) ≥80×109/L;
  2. Biochemical examination: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5×ULN; Serum total bilirubin (TBIL) ≤1.5×ULN; Serum creatinine (Cr) ≤1.5×ULN, or creatinine clearance ≥60mL/min;
  3. Coagulation function: activated partial thromboplastin time (APTT), International standardized ratio (INR), prothrombin time (PT) ≤1.5×ULN;
  4. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) ≥50%;
  5. Assessed with adequate organ function by doctors. 9. Fertile subjects must use appropriate methods of contraception during the study period and within 120 days after the end of the study, have a negative serological pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
3-year Disease-free survival (DFS) | UP to 3 years after surgery
  DFS is based on RECIST(Response Evaluation Criteria in Solid Tumours) 1.1 as assessed by the investigator and is defined as the time from surgery initiation to the date of first documentation of disease recurrence or death due to any cause

SECONDARY OUTCOMES:
major pathologic response (MPR) | an average of 2 to 4 weeks after surgery
  defined as the percentage of residual viable tumour cells in the tumour bed of no more than 10% after neoadjuvant therapy.
R0 resection rate | an average of 2 to 4 weeks after surgery
  defined as the absence of tumor cells present at the resection margin under microscope
Overall Survival (OS) | UP to 5 years after surgery
  defined as the time from randomization to death due to any cause.
Percentage of Participants Who Experience One or More Adverse Events (AEs) | Up to approximately 36 months
  An AE is based on NCI-CTC (The National Cancer Institute Common Toxicity Criteria) 5.0 as assessed by the investigator and is defined as any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The percentage of participants who experience at least one AE will be presented.
nutritional status | UP to 3 years after surgery
  Nutrition was assessed with the patient-generated subjective global assessment (PG-SGA).
quality of life | UP to 3 years after surgery
  Questionnaire includes EORTC QLQ-C30 (The European Organization for Reasearch and Treatment of Cancer Quality of Life Questionnare-Core 30))(version 3),

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR
Time Frame: partial data will be shared 3 years after the study was completed and end in 5 years.
Access Criteria: A shared data acquisition scheme approved by the researcher